CLINICAL TRIAL: NCT06635720
Title: REduced-dose Steroid PrOtocol for Childhood Nephrotic SyndromE (RESPONSE): a Pilot Open-label Randomized, Controlled Trial
Brief Title: REduced-dose Steroid PrOtocol for Childhood Nephrotic SyndromE (RESPONSE)
Acronym: RESPONSE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Rulan Parekh, Staff physician, clinician-scientist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000081679
Record Dates: First submitted 2024-09-30; First posted 2024-10-10 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Nephrotic Syndrome in Children; Nephrotic Syndrome, Minimal Change; Nephrotic Syndrome; Nephrotic Syndrome，Idiopathic
Keywords: Nephrotic syndrome; Idiopathic nephrotic syndrome; Childhood nephrotic syndrome; Minimal change disease; Focal segmental glomerulosclerosis
MeSH Terms: conditions — Nephrosis, Lipoid; Nephrotic Syndrome; Glomerulosclerosis, Focal Segmental | interventions — Prednisone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reduced-dose steroids (Experimental): Reduced-dose steroid protocol (intervention): oral prednisone or prednisolone 30mg/m2 (1mg/kg; max 40mg) daily until remission, then 20mg/m2 (0.66mg/kg; max 25mg) on alternate days for four weeks.
  Interventions: Drug: Prednisone
- Standard-dose steroids (Active Comparator): Standard-dose steroid protocol (control): oral prednisone or prednisolone 60mg/m2 (2mg/kg; max 60mg) daily until remission, then 40mg/m2 (1.5mg/kg; max 50mg) on alternate days for four weeks.
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — This study will compare two steroid dosing protocols for the treatment of childhood nephrotic syndrome relapses. The medications used for both intervention and control arms are oral prednisone 5mg tablets (DIN: 00312770) for children able to swallow or use crushed tablets, or oral prednisolone sodium phosphate 5mg base/5mL liquid (DIN: 02245532). Participants hospitalized after study enrollment will be permitted to switch to intravenous methylprednisolone sodium succinate (DIN: 02367955) at the same dose without being considered to have violated their treatment assignment.
  Other Names: Prednisolone

SUMMARY:
This is a pilot feasibility study for a proposed full-scale randomized controlled trial to evaluate the effectiveness and safety of a reduced-dose oral prednisone (steroids) regimen to treat childhood steroid-sensitive nephrotic syndrome relapses versus standard-dose prednisone (i.e., usual standard of care).

This internal pilot study is a single-center, open-label, randomized controlled trial at The Hospital for Sick Children (Toronto, ON, Canada). The primary objective of this pilot study is to determine the feasibility, safety, and resources needed to conduct the future full-scale randomized controlled trial.

DETAILED DESCRIPTION:
Study design:

This is a pilot study for a planned multi-center, Bayesian adaptive, non-inferiority RCT (Figure 1). This planned multi-center RCT will require additional funding, which we will apply for if feasibility is shown by this pilot. This pilot is a single-center (SickKids) open-label RCT comparing reduced vs. standard-dose steroids to treat nephrotic syndrome relapses.

Study population:

We will include children (1-18 years) from Ontario, Canada that are diagnosed with idiopathic SSNS and present in relapse (≥3+ dipstick protein or protein:creatinine ratio ≥200mg /mmol for ≥3 consecutive days). We will exclude children that have received >2 days of standard-dose prednisone; are on maintenance high-dose prednisone (>0.3mg/kg per day or >0.6mg/kg alternate days); have relapsed within the past 6 weeks; have grade 3+ peripheral edema (i.e., moderate-severe); are hospitalized; have stage 2+ acute kidney injury; or have thromboembolism. Children receiving other steroid-sparing immunosuppressives are eligible, but target drug levels will remain constant until the 2-week visit. No additional laboratory or imaging tests are needed, to maximize recruitment.

Interventions:

Reduced-dose steroids (intervention): oral prednisone 30mg/m2 (1mg/kg; max 40mg) daily until remission, then 20mg/m2 (0.66mg/kg; max 25mg) on alternate days for four weeks.

Standard-dose steroids (control): oral prednisone 60mg/m2 (2mg/kg; max 60mg) daily until remission, then 40mg/m2 (1.5mg/kg; max 50mg) on alternate days for four weeks.

Randomization 1:1 using permuted blocks. If a participant does not achieve remission by 2-weeks, develops symptomatic edema, stage 2+ acute kidney injury, or thromboembolism, they will be escalated to standard-dose steroids.

Outcomes:

The primary outcome is recruitment rate (number enrolled per month), since it is the greatest anticipated barrier to RCT feasibility. Other feasibility, tolerability, and safety outcomes are listed in Table 1. The pilot study will test case report forms, data management, quality control, and training systems. We will estimate treatment effect for the full-scale RCT's primary outcome (complete remission without steroid dose escalation by 2-weeks), to re-estimate sample size and evaluate full-scale RCT feasibility.

Sample size:

For this pilot study, we will recruit 50 children (25 per arm), which is 15% of the estimated sample size of the full-scale RCT. Sample size for this pilot must be adequate to assess RCT feasibility.

ELIGIBILITY:
Inclusion Criteria:

1. Provide informed consent ± assent
2. Participant age 1-18 years
3. Diagnosis of idiopathic nephrotic syndrome (defined as nephrotic-range proteinuria [first morning or 24-hour urine protein/creatinine ratio ≥200mg/mmol or ≥3+ protein on dipstick] and either hypoalbuminemia [serum albumin <30g/L] or edema)
4. Active nephrotic syndrome relapse at time of enrolment (defined as recurrence of nephrotic-range proteinuria [≥3+ protein on dipstick for ≥3 consecutive days18 OR first morning or 24-hour urine protein/creatinine ratio ≥200mg/mmol AND ≥1+ protein on dipstick for ≥3 consecutive days])
5. Ability to take oral medication and willingness to adhere to either study prednisone regimen
6. Ability and willingness to adhere to home urine and symptom monitoring during the initial two-week period after assigned treatment initiation
7. Have not been previously included in the RESPONSE trial
8. Participant located in Ontario, Canada at the time of study enrolment

Exclusion Criteria:

1. Prednisone treatment (at any dose) for the active relapse episode for >2-days prior to study enrolment
2. Relapse episode within the past 6-weeks (i.e., date of relapse onset within 6-weeks prior to date of enrolment)
3. Current receipt of high-dose maintenance prednisone therapy (dose >0.6mg/kg on alternate days or >0.3mg/kg daily)
4. Steroid-resistant nephrotic syndrome classification (defined as lack of complete remission within 6-weeks after initiating daily steroid treatment at a standard dose for the initial episode of nephrotic syndrome)
5. Congenital or monogenic cause of nephrotic syndrome (defined as age at diagnosis <1-year or known/suspected monogenic cause of nephrotic syndrome)
6. Secondary cause of nephrotic syndrome (includes membranous nephropathy, post-infectious glomerulonephritis [GN], complement-mediated GN [e.g., C3 glomerulopathy and immune complex-GN], IgA nephropathy, IgA vasculitis, lupus nephritis, medication-induced nephrotic syndrome, malignancy-induced nephrotic syndrome, active hepatitis B or C infection, or active HIV infection)
7. Presence of moderate-to-severe peripheral edema (grade 3+; indentation depth ≥5mm and rebound time >15 seconds)
8. Hospitalization since the onset of the active relapse episode
9. Acute kidney injury (KDIGO stage ≥1) since the onset of the active relapse episode
10. Active or prior known or suspected venous thromboembolism during a relapse episode
11. Active pregnancy or lactation
12. Any condition or diagnosis, that could in the opinion of the Principal Investigator or delegate interfere with the participant's ability to comply with study instructions, might confound the interpretation of the study results, or put the participant at risk

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Study recruitment rate | 1 year
  Number of participants enrolled per study month

SECONDARY OUTCOMES:
Treatment effect - treatment failure | From enrolment to 2-week study visit
  Failure to achieve complete remission or steroid dose escalation by 2-weeks
Number of eligible participants | 1 year
  Number (%) of screen eligible participants
Number of participants that initiate assigned treatment | 1 year
  Number (%) of participants that initiate assigned treatment
Participant drop-out rate | 1 year
  Number (%) of study participants that drop out
Treatment preference | 1 year
  Treatment preference ratings
Hospitalizations | From enrolment to 1 year
  Number (%) of participants that are hospitalized
Cumulative steroid dose | From enrolment to 1 year
  Cumulative steroid dose (mg/kg) prescribed
Adverse events | From enrolment to 1 year
  Number (%) of participants that experience adverse events and serious adverse events
Treatment adherence | From enrolment to 1 year
  Number (%) of participants that are adherent to assigned treatment and urine testing
Number of participants that complete 2-week study visit | 2 weeks
  Number (%) of participants that complete 2-week study visit

CONTACTS AND LOCATIONS:
Overall Officials: Rulan Parekh, MD MS, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No